CLINICAL TRIAL: NCT01233752
Title: Association Between Clinical Effect of Morphine in Patients With PCA After Major Surgery and Pharmacogenetics: Prospective Observational Clinical Study.
Brief Title: Association Between Clinical Effect of Morphine With PCA After Surgery and Pharmacogenetics
Acronym: PCA-Gene
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PT-SM-07-PCA-Gene
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Anesthesia; Surgery
Keywords: systemic morphine analgesia; pharmacogenetics; pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — genes OPRM1, COMT, UGTs, ESR1
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: Homozygous patients,using PCA administration with morphine chlorhydrate for postoperative analgesia, for the more frequent allele of the polymorphism A118G of OPRM1 gene
  Interventions: Drug: morphine chlorhydrate
- Group B: Both homozygous and heterozygous patients,using PCA administration with morphine chlorhydrate for postoperative analgesia, for the less frequent allele of the polymorphism A118G of OPRM1 gene
  Interventions: Drug: morphine chlorhydrate

INTERVENTIONS:
Drug: morphine chlorhydrate — The drug will be administrated by a bolus 45 minutes before the end of the surgery, with the following modalities: bolus with morphine chlorhydrate 0.15 mg/kg ± 20%. Also acetaminophene 1g and ketoprofen 160 mg (ketorolac 30mg) will be administrated during the operation.
  At the exit of the operative compartment patients will have an electronic pump (PCA) for 48h with morphine chlorhydrate to be used in boluses by 1 mg with a lock out of 5 mins, max dose 20 mg in 4 hours.
  Moreover, ketoprofen will be prescribed 160 mg x 2 per day (ketorolac 30mg x 2) (in case of allergy acetaminophene 1g x 3 daily).
  Postoperative analgesic treatment is lasting 48h for each patient (between starting of the PCA infusion (T0) and the following 48h).
  Other Names: morfina cloridrato

SUMMARY:
Identification of the genetic polymorphisms that could be correlated either with a better clinical response or with a major predisposition of patients to develop tolerance and/or side effects to the treatment with morphine.

DETAILED DESCRIPTION:
Valuation of the medium morphine dose (mg/kg/die) necessary to maintain NRS<4 in the first 24 hours post-surgery in the two groups of patients, A e B. Group A: homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene (about 80%); group B: both homozygous and heterozygous patients for the less frequent allele (about 20%).

In order to avoid the bias related to alterations in metabolism, patients with Cmax and AUC of morphine (and metabolites M6G and M3G) >2 standard deviation higher than expected population curve ("outliers") will be excluded for the primary purpose.

ELIGIBILITY:
Inclusion criteria:

* Males and females over 18 years, under 75 years, scheduled for postoperative pain control by PCA morphine administration
* HIV negative
* Classification American Society of Anesthesiologists (ASA) I: without systemic disease
* Classification ASA II or III (mild systemic disease or severe systemic disease that limits the activity without invalidity).
* Undergoing abdominal and urologic major surgery (neither urgent nor emergency surgery)
* Signed informed consent

Exclusion criteria:

* Usual assumption of analgesic opioids
* Cognitive alterations nor mental retardation
* Severe hepatic/renal insufficiency (cholinesterase <3000 mU/ml, total bilirubinaemia <2 mg/dl and creatininaemia <1.2 mg/dl)
* Inpatients in intensive therapy, either with sedation and/or mechanic ventilation.
* Allergies to morphine and derivates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pazients scheduled for major abdominal or urological surgery with postoperative pain control by PCA morphine administration
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the medium morphine dose (mg/kg/die)in the two groups homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene; group B: both homozygous and heterozygous patients for the less frequent allele | first 24 h after surgery
  Valutation of the medium morphine dose (mg/kg/die) necessary to maintain NRS<4 in the first 24 hours post-surgery in the two groups of patients, A e B. Group A: homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene (about 80%); group B: both homozygous and heterozygous patients for the less frequent allele (about 20%).

SECONDARY OUTCOMES:
Variants at the loci OPRM1, COMT, UGTs, ESR1,towards median pain measure | during 24 h postsurgery
  Frequency of the variants at the loci OPRM1, COMT, UGTs, ESR1, both in patients with NRS ≤4 and in those having NRS >4 at least once during 24 hours.
Detection of the medium morphine dose | First 24 h after surgery
  Detection of the medium morphine dose (mg/kg/die) necessary to maintain NRS<4 though the first 48 hours after surgery.
Pharmacokinetics of morphine with PCA after surgery | 48 h after surgery
  Pharmacokinetic study of both morphine and its principal active and/or toxic metabolites (M3G and M6G).
Variants frequency at loci OPRM1, COMT, UGTs, ESR1 | Within 48h after surgery
  Variants frequency at loci OPRM1, COMT, UGTs, ESR1 in the patients with Cmax and AUC of both morphine and M3G-M6G metabolites >2 standard deviations higher than expected population curve ("outliers").
Detection of the possible side effects. | 72 h postopratively
Detection of the association between M3G/M6G ratio and polymorphisms of UGTs (and possible side effects). | within 72 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Allegri, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (2):
- Italy (2):
  - Azienda Ospedaliera San Gerardo, Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia

REFERENCES:
- [Derived] Cattaneo S, Ingelmo P, Scudeller L, Gregori M, Bugada D, Baciarello M, Marchesini M, Alberio G, Normanno M, Jotti GS, Meschi T, Fanelli G, Massimo A. Sex differences in the daily rhythmicity of morphine consumption after major abdominal surgery. J Opioid Manag. 2017 Mar/Apr;13(2):85-94. doi: 10.5055/jom.2017.0372. PMID 28829523
- [Derived] De Gregori M, Diatchenko L, Ingelmo PM, Napolioni V, Klepstad P, Belfer I, Molinaro V, Garbin G, Ranzani GN, Alberio G, Normanno M, Lovisari F, Somaini M, Govoni S, Mura E, Bugada D, Niebel T, Zorzetto M, De Gregori S, Molinaro M, Fanelli G, Allegri M. Human Genetic Variability Contributes to Postoperative Morphine Consumption. J Pain. 2016 May;17(5):628-36. doi: 10.1016/j.jpain.2016.02.003. Epub 2016 Feb 21. PMID 26902643